CLINICAL TRIAL: NCT00017472
Title: Phase I Study of Thrice Weekly Hu1D10*in Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma and Acute Leukemia
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Chronic Lymphocytic Leukemia, Lymphocytic Lymphoma, Acute Lymphoblastic Leukemia, or Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01405; OSU 0101; OSU-0101; NCI-1254; OSU-00H0230; CDR0000068695; U01CA076576 (NIH)
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Splenic Marginal Zone Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Small Lymphocytic Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — apolizumab

ARMS (1):
- Arm I (Experimental): Patients receive apolizumab IV over at least 2 hours on days 1, 2, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with a complete or partial response who relapse after 2 months may receive an additional course of therapy provided they still express the 1D10 antigen.
  Interventions: Biological: apolizumab; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: apolizumab — Given IV
  Other Names: 1D1O Anti-lymphoma Antibody; MOAB 1D10; MoAb Hu1D10; Monoclonal antibody 1D10; Monoclonal Antibody Hu1D10
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have chronic lymphocytic leukemia, lymphocytic lymphoma, acute lymphoblastic leukemia, or acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) or biological effective dose of monoclonal antibody Hu1D10 (apolizumab) in patients with previously treated chronic lymphocytic leukemia or small lymphocytic lymphoma.

II. Determine the safety of this drug, in terms of frequency and severity of treatment-related adverse events, in this patient population.

SECONDARY OBJECTIVES:

I. Determine whether this drug has anti-leukemia/lymphoma activity in patients expressing the Hu1D10 antigen.

II. Determine the pharmacokinetics of this drug in this patient population. III. Determine whether the infusion-related toxicity of this drug is secondary to cytokine release in these patients.

IV. Determine whether the intensity of 1D10 target antigen on tumor cells is related to clinical response and treatment toxicity in these patients.

V. Determine the pharmacodynamics of this drug in this patient population.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to diagnosis (chronic lymphocytic leukemia or small lymphocytic lymphoma vs acute lymphoblastic leukemia [ALL] or acute myeloid leukemia [AML]). Patients with ALL or AML are enrolled after the maximum tolerated dose (MTD) is determined.

Patients receive apolizumab IV over at least 2 hours on days 1, 2, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with a complete or partial response who relapse after 2 months may receive an additional course of therapy provided they still express the 1D10 antigen.

Cohorts of 3-6 patients receive escalating doses of MOAB Hu1D10 until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity (DLT). If no DLT is observed, the biological effective dose (BED) is determined in the above cohorts. The BED is defined as the dose at which at least 4 of 6 patients experience an acceptable minimum trough level and clinical response. An additional 24 patients (12 per stratum) are treated at the MTD.

Patients are followed at 1 week, 1 and 2 months, and then every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 35 patients (12 per stratum) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* One of the following diagnoses:

  * Histologically confirmed chronic lymphocytic leukemia (CLL) or non-contiguous stage II or stage III-IV small lymphocytic lymphoma (SLL)

    * Previously treated with at least 1 form of chemotherapy or immunotherapy
  * Histologically confirmed acute lymphoblastic leukemia (enrolled after the maximum tolerated dose (MTD) is determined)

    * Must have failed 1 prior therapy
    * Ineligible for allogeneic stem cell transplantation
  * Histologically confirmed acute myeloid leukemia (enrolled after the MTD is determined)

    * Primary refractory or relapsed (within the past year) disease
    * Ineligible for potential curative therapy
* Express Hu1D10 antigen

  * Greater than 2 times the mean fluorescence intensity of the control by flow cytometry (blood or bone marrow cells) OR
  * Positive by immunohistochemical staining (lymph node)
* Presenting with one of the following indications for treatment unless early bone marrow transplantation is planned (CLL or SLL patients only):

  * Disease-related progressive symptoms
  * Progressively worsening anemia or thrombocytopenia
  * Progressively worsening lymphadenopathy
  * Massive splenomegaly or hypersplenism
  * Hyperlymphocytosis (WBC greater than 200,000/mm3) or lymphocyte doubling time less than 12 months
  * Marrow failure secondary to marrow infiltration by leukemia or lymphoma
* Performance status - ECOG 0-2
* At least 2 years
* See Disease Characteristics
* Platelet count at least 50,000/mm^3 (without transfusion)
* Bilirubin no greater than 3 mg/dL (unless elevated secondary to tumor)
* Creatinine no greater than 2.0 mg/dL
* No prior decompensated congestive heart failure, unstable angina, or myocardial infarction within the past 6 months not corrected by percutaneous transluminal coronary angioplasty or surgery
* No active infection requiring oral or IV antibiotics
* No other malignancy that would limit life expectancy
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study
* See Disease Characteristics
* At least 1 month since prior rituximab or alemtuzumab (unless CD20 or CD52 antigen is expressed on tumor cells)
* No prior monoclonal antibody Hu1D10
* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2001-04; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose level below which two or more of six patients experience a DLT assessed using NCI CTC version 2.0 | Up to 30 days

SECONDARY OUTCOMES:
Evaluation of the degree of apoptosis induced by ex vivo incubation of human CLL cells with Hu1D10 | Up to 1 year
  Descriptive data will be computed and compared using analysis of variance and non-parametric rank equivalents for continuous data and chi-square or Fisher's exact test for discrete data. Nevertheless, low statistical power will greatly limit these analyses.
Cytokine release | Up to 1 year
  Descriptive data will be computed and compared using analysis of variance and non-parametric rank equivalents for continuous data and chi-square or Fisher's exact test for discrete data. Nevertheless, low statistical power will greatly limit these analyses.
Caspase activation | Up to 1 year
  Descriptive data will be computed and compared using analysis of variance and non-parametric rank equivalents for continuous data and chi-square or Fisher's exact test for discrete data. Nevertheless, low statistical power will greatly limit these analyses.
Signaling and expression of apoptosis protein | Up to 1 year
  Descriptive data will be computed and compared using analysis of variance and non-parametric rank equivalents for continuous data and chi-square or Fisher's exact test for discrete data. Nevertheless, low statistical power will greatly limit these analyses.

CONTACTS AND LOCATIONS:
Overall Officials: John Byrd, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States